CLINICAL TRIAL: NCT02929017
Title: Integrating Palliative Care for Patients With Idiopathic Pulmonary Fibrosis and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kathleen O. Lindell, PhD, RN, Research Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO16070539; 1K23NR016276-01A1 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Fibrosis; IPF; Caregivers; Pulmonary; Palliative; end of life; Idiopathic
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis; Death | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Group will receive SUPPORT, an intervention that provides information about the disease, self-management strategies, and introduction to advanced care planning in a format with enhanced content available across multiple domains (face-to-face, printed material, and digitally (via use of a tablet) delivered by an interventionist.
  Interventions: Other: SUPPORT
- Usual Care (Other): Group will receive usual standard-of-care, and be provided with currently available printed material for information about their illness.
  Interventions: Other: Currently Available Printed Material

INTERVENTIONS:
Other: SUPPORT — Members of this group will receive personal, enhanced printed materials, as well as face-to-face support, and digital information provided by the interventionist.
  Arms: Intervention
Other: Currently Available Printed Material — Subjects will receive their usual standard of care, including currently available printed patient material.
  Other Names: Usual Standard of Care
  Arms: Usual Care

SUMMARY:
Patients with Idiopathic Pulmonary Fibrosis (IPF) and their caregivers will be randomized to receive this intervention or usual care. The intervention will include information about the disease, self-management strategies, and introduction to advanced care planning in a format with enhanced content available across multiple domains (face-to-face, printed material, digital (tablet) delivered by an interventionist. The usual care group will be provided with routine printed patient education.

At the end of life, IPF patients and their caregivers experience stress, symptom burden, poor quality of life, and inadequate preparedness for end-of-life care planning. The proposed study will measure feasibility, acceptability, and impact of a Supportive Care intervention.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis (IPF) is a disease of aging associated with intense medical and financial burden and expected to grow in incidence within the US population. Median survival from diagnosis is 3.8 years, although some patients succumb to a rapid death within 6 months. New therapies have recently become available. While these medications slow the rate of pulmonary deterioration, they have no impact on ultimate survival or quality of life. Although transplantation is an effective surgical therapy, less than 20% of patients ever receive a lung transplant. The remaining 80% have few treatment options and a likely rapidly progressive downhill course. Despite the fatal prognosis, we have found that patients and caregivers often fail to understand the poor prognosis as the disease relentlessly progresses. At the end of life, IPF patients and their caregivers experience stress, symptom burden, poor quality of life, and inadequate preparedness for end-of-life care planning.

The proposed study will measure feasibility, acceptability, and impact of a Supportive Care intervention. Patients with IPF and their caregivers will be randomized to receive this intervention or usual care. The intervention will include information about the disease, self-management strategies, and introduction to advanced care planning in a format with enhanced content available across multiple domains (face-to-face, printed material, digital (tablet) delivered by an interventionist. The usual care group will be provided with routine printed patient education.

ELIGIBILITY:
Inclusion Criteria:

* 45 years or older
* Primary Diagnosis of with Idiopathic Pulmonary Fibrosis (IPF)
* Has a caregiver, 18 years or older (spouse/partner/child/family member/friend), willing to participate.
* Sees a Simmons Center Physician for usual IPF care.

Exclusion Criteria:

* less than 45 years
* Not diagnosed with IPF
* Has an unwilling caregiver, or a caregiver under 18.
* Does not see a Simmons Center Physician for usual IPF care.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Stress | 3 years
  Perceived Stress Scale at baseline and completion of study in patients and caregivers

SECONDARY OUTCOMES:
Disease Preparedness | 3 years
  Survey to measure preparation for disease course at completion of study for patients and caregivers.
Knowledge | 3 years
  Survey to measure knowledge of IPF at baseline and study completion with patients and caregivers
Advance Care Planning | 3 years
  Survey to measure completion of advance care plan at study completion with patients
Quality of Dying and Death | 3 years
  Quality of Dying and Death for caregivers if patient deceased during study
Symptom Burden | 3 years
  Promis-29 to measure symptom burden in patients at baseline and study completion.
Health Related Quality of Life in IPF | 3 years
  ATAQ-IPF instrument to measure quality of life in patients at baseline and study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen O Lindell, PhD, RN, Principal Investigator — Dorothy P. and Richard P. Simmons Center for ILD
Locations (1):
- Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindell KO, Klein SJ, Veatch MS, Gibson KF, Kass DJ, Nouraie M, Rosenzweig MQ. Nurse-Led Palliative Care Clinical Trial Improves Knowledge and Preparedness in Caregivers of Patients with Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2021 Nov;18(11):1811-1821. doi: 10.1513/AnnalsATS.202012-1494OC. PMID 34003726
- [Derived] Lindell KO, Nouraie M, Klesen MJ, Klein S, Gibson KF, Kass DJ, Rosenzweig MQ. Randomised clinical trial of an early palliative care intervention (SUPPORT) for patients with idiopathic pulmonary fibrosis (IPF) and their caregivers: protocol and key design considerations. BMJ Open Respir Res. 2018 Feb 19;5(1):e000272. doi: 10.1136/bmjresp-2017-000272. eCollection 2018. PMID 29531748